CLINICAL TRIAL: NCT03709082
Title: A Phase I/II Study of Palbociclib, Letrozole and T-DM1 in Trastuzumab Refractory Estrogen Receptor Positive (ER+) and HER2 Positive Metastatic Breast Cancer
Brief Title: Palbociclib in Estrogen Receptor Positive (ER+) Human Epidermal Growth Factor Receptor 2 Positive (HER2+) Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Lauren Nye, Assistant Professor, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-IIT-HER2-Aspire
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: HER2-positive Breast Cancer; Breast Cancer Metastatic
Keywords: palbociclib
MeSH Terms: interventions — palbociclib; Letrozole; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Phase 1: Palbociclib 75 mg (Experimental): Palbociclib 75 milligrams (mg) by mouth (PO) daily Letrozole 2.5 mg PO Daily Ado-trastuzumab Emtansine (T-DM1) 3.6 milligrams per kilograms (mg/kg) intravenous (IV) Day 1
  Interventions: Drug: Palbociclib 75mg; Drug: Letrozole 2.5mg; Drug: T-DM1
- Phase 1: Palbociclib 100 mg (Experimental): Palbociclib 100 milligrams (mg) by mouth (PO) daily Letrozole 2.5 mg PO Daily Ado-trastuzumab Emtansine (T-DM1) 3.6 milligrams per kilograms (mg/kg) intravenous (IV) Day 1
  Interventions: Drug: Letrozole 2.5mg; Drug: T-DM1; Drug: Palbociclib 100mg
- Phase 1: Palbociclib 125 mg (Experimental): Palbociclib 125 milligrams (mg) by mouth (PO) daily Letrozole 2.5 mg PO Daily Ado-trastuzumab Emtansine (T-DM1) 3.6 milligrams per kilograms (mg/kg) intravenous (IV) Day 1
  Interventions: Drug: Letrozole 2.5mg; Drug: T-DM1; Drug: Palbociclib 125mg
- Phase 2: RP2D (Experimental): Recommended Phase 2 dose (RP2D; determined during Phase 1 Safety Run In) Palbociclib by mouth (PO) daily Letrozole 2.5 mg PO Daily Ado-trastuzumab Emtansine (T-DM1) 3.6 milligrams per kilograms (mg/kg) intravenous (IV) Day 1
  Interventions: Drug: Letrozole 2.5mg; Drug: T-DM1; Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib 75mg — Oral Administration
  Other Names: Ibrance
  Arms: Phase 1: Palbociclib 75 mg
Drug: Letrozole 2.5mg — Oral Adminstration
  Other Names: Femara
Drug: T-DM1 — Intravenous Administration
  Other Names: Ado-trastuzumab Emtansine; Kadcyla
Drug: Palbociclib 100mg — Oral Administration
  Other Names: Ibrance
  Arms: Phase 1: Palbociclib 100 mg
Drug: Palbociclib 125mg — Oral Administration
  Other Names: Ibrance
  Arms: Phase 1: Palbociclib 125 mg
Drug: Palbociclib — Oral Administration
  Other Names: Ibrance
  Arms: Phase 2: RP2D

SUMMARY:
This study will determine the recommend dose of palbociclib in combination with letrozole and another medication, Ado-trastuzumab emtansine (T-DM1). Additionally, researchers will determine how well this recommended dose will improve outcomes in this type of advanced breast cancer.

The study will include a safety lead-in with escalating dosing of palbociclib to determine the recommended phase II dose (RP2D) of palbociclib in this combination and an expanded phase II of palbociclib at the RP2D in combination with letrozole and Ado- trastuzumab Emtansine (T-DM1).

The starting dose of palbociclib will be 75 milligrams (mg) by mouth (PO) daily for each 21 day cycle. If 0 of 3 patients at the 75mg dose level experience a dose limiting toxicity (DLT), the next 3 patients will be enrolled at the next higher dosing cohort of 100mg PO daily for each 21 day cycle. If 0 of 3 patients at the 100mg dose level experience a DLT, the next 3 patients will be enrolled at the next higher dosing cohort of 125mg PO daily for each 21 day cycle. If 0 of 3 patients at the 125mg dose level experience a DLT, 125mg PO daily of palbociclib will be the phase II recommended dose used in the phase II expanded cohort. Patients receiving the phase II recommended dose in phase I will be enrolled in phase II of the study.

During safety lead-in and expanded phase II, Letrozole 2.5mg PO will be administered daily for each 21 day cycle and T-DM1 3.6 milligrams per kilograms intravenously (IV) will be administered on Day 1 of each 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of Estrogen Receptor (ER) positive and HER2 (human epidermal growth factor receptor 2) positive metastatic breast cancer based on local laboratory results.
* Prior treatment with a taxane (including paclitaxel, docetaxel and/or nanoparticle protein-bound paclitaxel).
* Prior treatment with trastuzumab with or without pertuzumab.
* Measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
* Eastern Cooperative Oncology Group Performance Status of 0-2
* Adequate organ and marrow function
* Women must be post-menopausal
* Must be able to swallow pills

Exclusion Criteria:

* Current or anticipated use of other investigational agents
* Prior therapy with a cyclin-dependent kinase 4/6 inhibitor
* Subject has received chemotherapy or radiotherapy within 14 days prior to Cycle 1, Day 1 of the study or has not recovered from adverse events due to agents administered more than 14 days earlier
* Subject has leptomeningeal disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib or other agents used in study
* Subject has other illness or disease that the investigator believes will interfere with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Rate of Overall Response | From the time of first documented complete response or appearance of one or more new lesions, until the first documented date of recurrent or progressive disease, whichever came first, assessed up to 5 years
  Determine overall response rate (ORR), defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Proportion of participants with complete response (CR). | Up to 5 years
  Defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Proportion of participants with partial response (PR). | Up to 5 years
  Defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Proportion of participants with stable disease (SD). | Up to 5 years
  Defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Proportion of participants with Grade 3 or higher adverse event. | Up to 5 years
  Defined per Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Number of patients with adverse events | Up to 5 years
  Determine safety and tolerability of the intervention, defined per Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Number of participants with a worsening Patient Reported Outcomes of Adverse Events (PRO-AE) score | At baseline and Day 1 of each cycle, up to 5 years (each cyle is 21 days)
  PRO-AE score defined per Patient Reported Outcome Measurement Information System (PROMIS) and Breast Cancer Prevention Trial (BCPT) Symptom Checklist.
Peak observed plasma concentration | Cycle 1, Day 1: 0 ,2,4 and 8 hours post treatment; Cycle 1, Day 15: 0 hours post treatment (each cyle is 21 days)
  Defined per maximum observed concentration (Cmax) and time of Cmax (Tmax).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Nye, MD, Principal Investigator — KUCC
Locations (5):
- United States (5):
  - The University of Kansas Cancer Center, West Clinic, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park Clinic, Overland Park, Kansas
  - The University of Kansas Cancer Center, North Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit Clinic, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No